CLINICAL TRIAL: NCT07045532
Title: Assessment the Effectiveness of Bronchoscopic Thermal Vapor Ablation in Chronic Obstructive Pulmonary Disease and Ablation in Pulmonary Nodules by Pulmonary Magnetic Resonance Imaging
Brief Title: Assessment the Effectiveness of BTVA in COPD and Ablation in Pulmonary Nodules by Pulmonary MRI
Status: Recruiting | Type: Observational
Sponsor: Shanghai Chest Hospital (Other)
Responsible Party: Principal Investigator, Jiayuan Sun, Vice dean of the hospital, Shanghai Chest Hospital
Other Study IDs: KS(Y)23216
Record Dates: First submitted 2025-06-04; First posted 2025-07-01 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2024-09

CONDITIONS: COPD; Lung Cancers
Keywords: MRI; COPD; Lung cancer; ablation
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive; Lung Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A Clinical Study Based on Magnetic Resonance Imaging of the Lungs to Assess the Efficacy of Thermal Vapor Ablation and Pulmonary Nodule Ablation in Chronic Obstructive Pulmonary Disease After Surgery.

The efficacy of hot steam ablation for chronic obstructive pulmonary disease was evaluated using the innovative MRI sequence PREFUL_MRI, and the efficacy of pulmonary nodule ablation was evaluated using the innovative MRI sequence GRASP_MRI.

ELIGIBILITY:
Inclusion Criteria:

1. Age >18 years old;
2. Patients with pulmonary nodules: patients with pulmonary nodules indicated by chest CT, pathologically diagnosed as malignant, and receiving ablative treatment, including transthoracic and percutaneous ablative methods, including radiofrequency, microwave, and freezing;
3. COPD patients: patients diagnosed with COPD according to the GOLD principle and treated with thermal steam ablation for COPD;
4. Understand the study and sign the informed consent.

Exclusion Criteria:

1. Chest CT nodules in patients with pulmonary nodules were pure ground glass nodules;
2. Patients who install or carry metal implants such as cardiac pacemakers, heart stents, artificial heart valves in the body or suffer from claustrophobia, allergy to contrast media and other reasons are not suitable for MRI examination;
3. severe cardiopulmonary dysfunction and other diseases that may significantly increase the risk of ablation surgery;
4. Patients with severe COPD exacerbation or pneumonia in the past four weeks;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients older than 18 years of age with pulmonary nodules and COPD.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-09-01 (Actual); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
PREFUL-MRI Ventilation and Perfusion Parameters in Patients with COPD Following Lung Volume Reduction Surgery with Thermal Steam | From enrollment to 6 months post-surgery
  Using the Phase-Resolved Functional Lung(PREFUL)-MRI dedicated post-processing analysis software, we can obtain images of the patient's lung ventilation and perfusion status.
PREFUL-MRI Ventilation and Perfusion Parameters in Patients with COPD Following Lung Volume Reduction Surgery with Thermal Steam | From enrollment to 6 months post-surgery
  Percentage of perfusion defect (QDP)：Calculation of QDP based on PREFUL-MRI dedicated post-processing software
PREFUL-MRI Ventilation and Perfusion Parameters in Patients with COPD Following Lung Volume Reduction Surgery with Thermal Steam | From enrollment to 6 months post-surgery
  Percentage of ventilation defect (VDP)：Calculation of VDP based on PREFUL-MRI dedicated post-processing software
PREFUL-MRI Ventilation and Perfusion Parameters in Patients with COPD Following Lung Volume Reduction Surgery with Thermal Steam | From enrollment to 6 months post-surgery
  Percentage of ventilation-perfusion match (VQM):Calculation of VQM based on PREFUL-MRI dedicated post-processing software
Quantitative Hemodynamic Analysis Parameters Based on Tofts Model Using GRASP-MRI After Ablation of Solid Pulmonary Nodules | From enrollment to 3 months post-surgery
  Quantitative parameters of GRASP-MRI images based on the Tofts model:
  Volume transfer coefficient(Ktrans)(/min)：the rate transfer constant of gadolinium between plasma and tissue interstitium;
Quantitative Hemodynamic Analysis Parameters Based on Tofts Model Using GRASP-MRI After Ablation of Solid Pulmonary Nodules | From enrollment to 3 months post-surgery
  Quantitative parameters of GRASP-MRI images based on the Tofts model:
  Interstitial volume(Ve)(0～1)：the extracellular-extravascular volume;
Quantitative Hemodynamic Analysis Parameters Based on Tofts Model Using GRASP-MRI After Ablation of Solid Pulmonary Nodules | From enrollment to 3 months post-surgery
  Quantitative parameters of GRASP-MRI images based on the Tofts model:
  Kep: Backflow rate constant, reflecting the time constant for returning from EES to the vascular system, Kep = Ktrans / Ve.

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai chest hospital, Shanghai, Shanghai Municipality, China